CLINICAL TRIAL: NCT03513692
Title: A Randomised Controlled Trial to Compare Post-operative Sensitivity of Restorations Completed With Fill-Up, a Dual Curing Composite and Conventional Composite Resin
Brief Title: A RCT to Compare Post-operative Sensitivity of Restorations With Fill-Up, a Dual Curing Composite and Conventional Composite Resin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, T Paul Hyde, Clinical Associate Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS project ID: 213486
Record Dates: First submitted 2018-04-18; First posted 2018-05-01 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Sensitivity of Existing Dental Filling Materials

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fill-Up composite resin (Active Comparator): In this arm of the study, participants will have the dental restoration completed with "FillUp" from Coltene, a composite resin a CE marked and licensed restorative material.
  Interventions: Device: Fill-Up composite resin
- Conventional; composite (Active Comparator): In this arm of the study, participants will have the dental restoration completed with a conventional composite resin using a CE marked and licensed restorative material.
  Interventions: Device: Fill-Up composite resin

INTERVENTIONS:
Device: Fill-Up composite resin — 2 arm study comparing restoration of a tooth with either FillUp composite or conventional composite
  Other Names: conventional composite resin

SUMMARY:
The trial compares patient-reported postoperative sensitivity of 2 existing dental filling materials. The dental filling materials will be used according to manufacturer's instructions and within the existing CE marked licence. We are interested in investigating which licensed material confers the least postoperative discomfort to our patients in normal clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is over 18
2. Patient is under 70
3. Patient is capable of informed consent
4. The tooth responds to sensitivity testing ('vitality test' with an electric pulp tester)
5. The cavity is suitable for composite restoration
6. The patient prefers composite to amalgam.
7. The restoration required involves 2 or more surfaces of the tooth

Exclusion Criteria:

1. The tooth does not respond to an electric pulp test
2. The patient is suffering dental pain at the time of consent
3. The patient is currently taking long term analgesics
4. The patient is incapable of giving informed consent
5. The patient is a child under 18
6. The patient is unable to return the VAS assessment sheets at the appropriate time
7. The tooth to be filled is periodontally involved (grade 2 or grade 3 mobile)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Post operative sensitivity | 1 month
  patient assessment by VAS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided